CLINICAL TRIAL: NCT02795325
Title: A Phase 1 Study of DCR-PH1 in Patients With Primary Hyperoxaluria Type 1 (PH1)
Brief Title: A Study of DCR-PH1 in Patients With Primary Hyperoxaluria Type 1 (PH1)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Dicerna Pharmaceuticals, Inc., a Novo Nordisk company (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCR-PH1-101
Record Dates: First submitted 2016-05-18; First posted 2016-06-10 (Estimated); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Primary Hyperoxaluria Type 1
Keywords: Primary Hyperoxaluria Type 1; PH1; Calcium Oxalate Stones; Kidney Stones; Liver Enzyme Deficiency; Genetic Diseases; Inborn Kidney Diseases; Metabolic Diseases; Inborn Errors; Urological Diseases; Carbohydrate Metabolism; Hyperoxaluria; AGT; RNAi; siRNA; DCR-PH1
MeSH Terms: conditions — Primary hyperoxaluria type 1; Kidney Calculi; Genetic Diseases, Inborn; Metabolic Diseases; Urologic Diseases; Hyperoxaluria

ARMS (2):
- PH Patients (Experimental)
  Interventions: Drug: DCR-PH1
- Healthy Volunteers (Experimental)
  Interventions: Drug: DCR-PH1; Other: Placebo

INTERVENTIONS:
Drug: DCR-PH1 — IV infusion of DCR-PH1
Other: Placebo
  Arms: Healthy Volunteers

SUMMARY:
A phase 1 study of DCR-PH1 in patients with primary hyperoxaluria type 1 (PH1) to determine the safety, tolerability, pharmacokinetic (PK) and pharmacodynamics (PD) effects of DCR-PH1 administered via-intravenous infusion (IV)

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 12 years of age
* Diagnosis of PH1, confirmed by genotyping
* 24-hour urine oxalate excretion as defined in the protocol
* eGFR ≥ 40 mL/min normalized to 1.73 m2 BSA
* Written informed consent for adults (≥18 years old, or per local regulatory requirement); written informed assent for adolescents (12 to <18 years old, or per local regulatory requirement)

Exclusion Criteria:

* Prior renal and/or hepatic transplantation
* Participation in any clinical study involving administration of any investigational drug within the 30 days before enrollment
* Pregnancy or lactation at the time of screening or enrollment
* Women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding and must be willing to use contraception
* Patients with a known history of human immunodeficiency virus (HIV) or active infection with hepatitis B virus or hepatitis C virus
* Moderate to severe liver impairment
* Liver function test abnormalities: alanine transaminases (ALT) and/or aspartate transaminases (AST) > 2 times upper limit of normal (ULN)
* History of severe reaction to a liposomal product or a known hypersensitivity to lipid products.
* Unable to collect required study samples or follow study procedures
* No clinically significant health concerns

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-05-13 (Actual); Primary Completion 2016-10-14 (Actual); Study Completion 2016-10-14 (Actual)

PRIMARY OUTCOMES:
The safety of DCR-PH1 evaluated by the proportion of subjects that experience adverse events (AEs) | Through Day 29

SECONDARY OUTCOMES:
Profile of pharmacokinetics (PK) of DCR-PH1 - Cmax | Through Day 29
Profile of pharmacokinetics (PK) of DCR-PH1 - tmax | Through Day 29
Profile of pharmacokinetics (PK) of DCR-PH1 - AUC | Through Day 29
Profile of pharmacokinetics (PK) of DCR-PH1 - t½ | Through Day 29
The effect of DCR-PH1 on plasma glycolate levels | Through Day 29
The effect of DCR-PH1 on urine glycolate levels | Through Day 29
The effect of DCR-PH1 on plasma oxalate levels | Through Day 29
The effect of DCR-PH1 on urine oxalate levels | Through Day 29

CONTACTS AND LOCATIONS:
Locations (2):
- Bonn, Germany
- Amsterdam, Netherlands

REFERENCES:
- [Background] Martin-Higueras C, Luis-Lima S, Salido E. Glycolate Oxidase Is a Safe and Efficient Target for Substrate Reduction Therapy in a Mouse Model of Primary Hyperoxaluria Type I. Mol Ther. 2016 Apr;24(4):719-25. doi: 10.1038/mt.2015.224. Epub 2015 Dec 22. PMID 26689264
- [Background] Milliner DS. siRNA Therapeutics for Primary Hyperoxaluria: A Beginning. Mol Ther. 2016 Apr;24(4):666-7. doi: 10.1038/mt.2016.50. No abstract available. PMID 27081720
- [Background] Dutta C, Avitahl-Curtis N, Pursell N, Larsson Cohen M, Holmes B, Diwanji R, Zhou W, Apponi L, Koser M, Ying B, Chen D, Shui X, Saxena U, Cyr WA, Shah A, Nazef N, Wang W, Abrams M, Dudek H, Salido E, Brown BD, Lai C. Inhibition of Glycolate Oxidase With Dicer-substrate siRNA Reduces Calcium Oxalate Deposition in a Mouse Model of Primary Hyperoxaluria Type 1. Mol Ther. 2016 Apr;24(4):770-8. doi: 10.1038/mt.2016.4. Epub 2016 Jan 13. PMID 26758691
- See also: Related Info — http://www.dicerna.com
- See also: Related Info — http://www.rarekidneystones.org
- See also: Related Info — http://www.ohf.org
- See also: Related Info — http://www.nord.org